CLINICAL TRIAL: NCT04770610
Title: A Phase III, Randomized, Double-masked, Placebo-controlled, Parallel-group, Multicenter Study of the Safety and Efficacy of OT-101 (Atropine Sulfate 0.01%) in Treating the Progression of Myopia in Pediatric Subjects
Brief Title: Study of OT-101 in Treating Myopia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocumension (Hong Kong) Limited (Other)
Collaborators: ORA, Inc. (Industry); Statistics & Data Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OT_101_001
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OT-101 alone (Experimental): Atropine Sulfate 0.01% Ophthalmic Solution through year 4
  Interventions: Drug: OT-101 Ophthalmic Solution
- OT-101 plus vehicle (Experimental): Atropine Sulfate 0.01% Ophthalmic Solution through year 3 followed by vehicle for 1 year
  Interventions: Drug: OT-101 Ophthalmic Solution; Drug: Vehicle
- Vehicle (Placebo Comparator): Vehicle (Investigational Product minus active ingredient) through year 4
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OT-101 Ophthalmic Solution — Atropine 0.01%
  Other Names: Investigational Product
  Arms: OT-101 alone; OT-101 plus vehicle
Drug: Vehicle — Investigational Product minus active ingredient
  Other Names: Placebo
  Arms: OT-101 plus vehicle; Vehicle

SUMMARY:
This is a phase III, randomized, double-masked, placebo-controlled, parallel-group, multicenter safety, tolerability, and efficacy study of atropine sulfate 0.01% (OT-101) as an investigational treatment for myopia in pediatric subjects

DETAILED DESCRIPTION:
This is a phase III, randomized, double-masked, placebo-controlled, parallel-group, multi-center study to evaluate the safety tolerability and efficacy of OT-101 (Atropine 0.01%) Ophthalmic Solution in treating the progression of myopia in pediatric subjects that will enroll approximately 678 pediatric subjects with myopia in total. Subjects will be stratified by age and refractive error.

This study consists of 11 visits over the course of approximately 4 years and can be broken down in the 3 stages: Screening (Days -14 to -1), Stage 1 (Day 1 to Year 3), and Stage 2 (Year 3 to Year 4). In stage 1, subjects will be randomized in a 2:1 manner to OT-101 Ophthalmic Solution: Placebo. Subjects will be dosed with one drop of study treatment per eye once daily at bedtime for 3 years. In stage 2, subjects will be re-randomization 1:1 will occur at Visit 9 (Month 36). At re-randomization, subjects who had been assigned to OT-101 Ophthalmic Solution will be randomized in a 1:1 ratio to continue on OT-101 Ophthalmic Solution or switch to placebo. Subjects who had been assigned to placebo will continue with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have refractive error by cycloplegic autorefraction at baseline (Visit 1) in the study eye of:

  1. myopia greater or equal to -1.00D of spherical equivalent
  2. astigmatism less than or equal to 1.50DC
  3. progression of at least -0.50D of spherical equivalent in the last 12 months;

     Exclusion Criteria:
* Have active or a history of chronic or recurrent episodes of ocular inflammation (e.g. moderate to severe blepharitis, allergic conjunctivitis, peripheral ulcerative keratitis, scleritis) in either eye;
* Have undergone any myopia control treatment including orthokeratology, rigid gas-permeable contact lenses, bifocal contact lenses, progressive addition spectacle lenses, or other lenses to reduce myopia progression in the previous 6 months. Myopic correction in the form of single-vision eyeglasses and/or single-vision soft contact lenses are allowed;
* Have undergone any form of refractive eye surgery including incisional keratotomy, photorefractive keratectomy [PRK], laser in situ keratomileusis [LASIK], laser-assisted sub- epithelial keratectomy [LASEK]), corneal inlay procedures, conductive keratoplasty, small incision lenticule extraction (SMILE), cataract extraction, or any form of intraocular lens implantation;

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 678 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of study eyes with a -0.75D of progressive myopia defined as an increase in spherical equivalent of -0.75D or greater as assessed by cycloplegic autorefraction. | At month 36
  Efficacy of OT-101 Ophthalmic Solution

SECONDARY OUTCOMES:
Change in spherical equivalent (D) in the study eye as assessed by cycloplegic autorefraction | Baseline to Month 36
  Efficacy of OT-101 Ophthalmic Solution
Change in study eye axial length as measured by cycloplegic biometry (a standardized device will be selected for this study) | Baseline to Month 36
  Efficacy of OT-101 Ophthalmic Solution

CONTACTS AND LOCATIONS:
Overall Officials: Keith Lane, Study Director — ORA, Inc.
Locations (15):
- United States (15):
  - Colorado Vision Institute, Colorado Springs, Colorado
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Family Focus, Gainesville, Florida
  - Pediatric Eye Consultants of North Florida, Jacksonville, Florida
  - Indiana University Health Physicians Pediatric Ophthalmology, Indianapolis, Indiana
  - Kids Eye Care of Maryland, Rockville, Maryland
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Pure Ophthalmic Research, Mint Hill, North Carolina
  - CORE, Inc., Shelby, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Scott & Christie and Associates, Cranberry Township, Pennsylvania
  - Pediatric Ophthalmology of Erie, Inc, Erie, Pennsylvania
  - UPMC Children's Hospital, Pittsburgh, Pennsylvania
  - Total Eye Care, P.A., Memphis, Tennessee
  - San Antonio Eye Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No